CLINICAL TRIAL: NCT07052630
Title: Improving Goals of Care Conversations With Hematopoietic Cell Transplant Survivors (IMPACT - HCT)
Brief Title: Patient Navigation and the Planning Advance Care Together Website to Improve Goals of Care Conversations in Hematopoietic Cell Transplant Survivors, IMPACT-HCT Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1125595; NCI-2025-04134 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20855 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-06-24; First posted 2025-07-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Patient Navigation; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1 (PACT, patient navigation) (Experimental): Patients interact with the PACT website over 4 weeks and receive a navigation session over 30-45 minutes with a trained health coach to review ACP.
  Interventions: Other: Internet-Based Intervention; Behavioral: Patient Navigation; Other: Survey Administration
- Condition 2 (patient navigation) (Experimental): Patients receive a navigation session over 30-45 minutes with a trained health coach to review ACP.
  Interventions: Behavioral: Patient Navigation; Other: Survey Administration
- Condition 3 (PACT) (Experimental): Patients interact with the PACT website over 4 weeks.
  Interventions: Other: Internet-Based Intervention; Other: Survey Administration
- Condition 4 (standard/usual care) (Active Comparator): Patients receive standard/usual care for 4 weeks on study.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Interact with PACT website
  Arms: Condition 1 (PACT, patient navigation); Condition 3 (PACT)
Behavioral: Patient Navigation — Receive a patient navigation session
  Other Names: Patient Navigator Program
  Arms: Condition 1 (PACT, patient navigation); Condition 2 (patient navigation)
Other: Best Practice — Receive standard/usual care
  Other Names: standard of care; standard therapy
  Arms: Condition 4 (standard/usual care)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the impact of patient navigation and the Planning Advance Care Together (PACT) website, either alone or in combination with one another, on advanced care planning (ACP) in patients with blood cancers who received a hematopoietic cell transplant (HCT). Engagement in ACP, including having goals of care conversations, improves quality of care at the end of life and supporting this should be included in all cancer survivorship care. Patient navigation is a healthcare service that is designed to guide a patient through the healthcare system and reduce barriers to timely screening follow-up, diagnosis, treatment, and supportive care. PACT is a web-based tool that provides information about ACP, assistance with documents for advanced directives, a supportive network and a forum for discussions about ACP. Patients who engage in ACP are more likely to have higher quality of life at the end of life, receive the care they want, die where they prefer, utilize hospice effectively, and are less likely to receive futile, aggressive care at the end of life. For HCT survivors at ongoing risk of death and other disease-related complications, having a plan in place for care they want is critical. Patient navigation and/or the PACT website may improve ACP, including completion of advance care directives and goals of care conversations, in patients with blood cancers who received an HCT.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 4 conditions.

CONDITION 1 (PACT + PATIENT NAVIGATION): Patients interact with the PACT website over 4 weeks and receive a navigation session over 30-45 minutes with a trained health coach to review ACP.

CONDITION 2 (PATIENT NAVIGATION ONLY): Patients receive a navigation session over 30-45 minutes with a trained health coach to review ACP.

CONDITION 3 (PACT ONLY): Patients interact with the PACT website over 4 weeks.

CONDITION 4 (NO PACT/NO PATIENT NAVIGATION): Patients receive standard/usual care for 4 weeks on study.

After completion of study intervention, patients are followed up at 4 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Received a transplant for a hematologic malignancy
* Current age 18 years of age or older
* Currently 1 to 5 years after HCT
* Ability to speak and read English
* Has not completed all advance directives and/or had a goals of care (GOC) conversation with their physician
* Access to the internet (via computer, tablet, or mobile device)

Exclusion Criteria:

* Unable to provide informed consent
* Uncontrolled psychiatric conditions (confirmed through electronic health record [EHR] by study staff)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Rate of enrollment) | At baseline
  Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data. Feasibility cutoffs will be based on prior research and include >= 50% of eligible patients will enroll in the study.
Feasibility (Rate of completion of intervention components) | At 12 weeks post intervention
  For the patient navigation component, this means that patients participate in the single patient navigation session with a health coach. For the Planning Advance Care Together (PACT) condition, this means that patients set up an account with the PACT website and engage in at least accessing the website. Feasibility cutoffs will be based on prior research and include >= 50% of enrolled patients will adhere to and complete assigned intervention components and study-related assessments.
Feasibility (Rate of completion of study assessments) | At baseline, and at 4 and 12 weeks post intervention
  Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data. Feasibility cutoffs will be based on prior research and include >= 50% of enrolled patients will adhere to and complete assigned intervention components and study-related assessments.
Acceptability of intervention | At 4 weeks post intervention
  Will be measured using the 4-item Acceptability of Intervention Measure. Items are rated on a 5-point Likert scale. Acceptability will be defined as a median score of >= 4.
Completion of advance directives | At baseline, and at 4 and 12 weeks post intervention
  Questions asking patients whether they have completed a do not resuscitate (DNR) order, living will or identified a health care proxy. This item is scored as having no advance directives (0) to all advance directives completed (3). In addition to the primary outcome of advance directives (0 to 3 score), investigators will also examine each outcome separately (e.g., yes/no to completing a health care proxy) as secondary measures.

SECONDARY OUTCOMES:
Discussion of advance care planning (ACP)/goals of care conversation | At baseline, and at 4 and 12 weeks post intervention
  Will be measured using the 8-item measure of discussing end-of-life care, living will, health care proxy and do not resuscitate (DNR) orders with family and doctor. Will be evaluated using a linear mixed model with effect coding.
Level of engagement in ACP | At baseline, and at 4 and 12 weeks post intervention
  Will be measured using the reliable and valid Advance Care Planning Engagement Survey: Action Measures. It is an 18-item measure assessing domains of decision maker, quality of life, flexibility, and asking questions about treatment and ACP (yes/no). Will be evaluated using a linear mixed model with effect coding.
Readiness to engage in ACP | At baseline, and at 4 and 12 weeks post intervention
  Will be assessed using a previously developed and validated questionnaire, the Advance Care Planning Readiness Scale. This is an 8-item questionnaire that asks questions about patients' readiness to engage in ACP on a 7-point Likert scale (1 = Strongly disagree, 7 = Strongly agree). Will be evaluated using a linear mixed model with effect coding.
Self-efficacy for treatment decision-making | At baseline, and at 4 and 12 weeks post intervention
  Will be measured by the Decision-Making Participation Self-Efficacy (DEPS) scale. The DEPS scale is a 5-item validated measure that assesses cancer patients' confidence in engaging in different activities related to decision-making. Patients are asked to indicate how confident they are that they would be able to engage in various decision-making activities (e.g., "Tell your doctor about the option you would prefer"); items are rated on a 5-point Likert scale (1 = not at all confident, 5 = completely confident). Will be evaluated using a linear mixed model with effect coding.
Psychological distress | At baseline, and at 4 and 12 weeks post intervention
  Will be measured using the Patient Health Questionnaire, an 8-item questionnaire assessing depression on a 4-point Likert scale (0 = not at all, 3 = nearly every day). Will be evaluated using a linear mixed model with effect coding.
Engagement with PACT website | At baseline, and at 4 and 12 weeks post intervention
  Will be assessed by capturing data to indicate the engagement levels with the PACT website for those randomly assigned to this component, including: number and frequency of visits to the website and time spent on each component of the website.
Engagement with patient navigation intervention (Completion rates of patient navigation intervention session) | At 4 weeks post intervention
  Will assess engagement with the patient navigation component for those randomly assigned to this component by tracking completion rates of the single, one time patient navigation session.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Shen, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No